CLINICAL TRIAL: NCT00107978
Title: A Phase 3, Randomized, Double-Blind, Multinational Trial of Intravenous Telavancin Versus Vancomycin for Treatment of Complicated Gram Positive Skin and Skin Structure Infections With a Focus on Patients With Infections Due to Methicillin-resistant Staphylococcus Aureus
Brief Title: Comparison of Telavancin and Vancomycin for Complicated Skin and Skin Structure Infections With a Focus on Methicillin-resistant Staphylococcus Aureus
Acronym: ATLAS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Steven Barriere, Pharm.D., Vice President, Clinical and Medical Affairs, Theravance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0018
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Staphylococcal Skin Infection
Keywords: cSSSI (complicated Skin and Skin Structure Infections); Staph (Staphylococcus); MRSA (Methicillin-resistant Staphylococcus Aureus)
MeSH Terms: conditions — Staphylococcal Skin Infections; Staphylococcal Infections | interventions — telavancin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telavancin (Experimental)
  Interventions: Drug: Telavancin
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Telavancin — Telavancin 10 mg/kg/day, IV for up to 14 days.
  Other Names: VIBATIV; TD-6424
  Arms: Telavancin
Drug: Vancomycin — Vancomycin 1 Gm IV administered every 12 hrs for up to 14 days.
  Arms: Vancomycin

SUMMARY:
Study 0018 (NCT00107978) compares the safety and effectiveness of an investigational drug, telavancin, and an approved drug, vancomycin, for the treatment of complicated skin and skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of one of the following complicated skin and skin structure infections with MRSA (Methicillin-resistant Staphylococcus Aureus) either suspected or confirmed as the major cause of the infection:

  * major abscess requiring surgical incision and drainage;
  * infected burn (see exclusion criteria for important qualifications);
  * deep/extensive cellulitis;
  * infected ulcer (see exclusion criteria for important qualifications);
  * wound infections
* Patients must be expected to require at least 7 days of intravenous antibiotic treatment.

Exclusion Criteria:

* Received more than 24 hours of potentially effective systemic (IV/IM or PO) antibiotic therapy
* Burns involving > 20% of body surface area or third degree/full thickness in nature, diabetic foot ulcers, ischemic ulcers/wounds, necrotizing fasciitis, gas gangrene, or mediastinitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2005-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke University
Locations (1):
- Louisiana State University Health Sciences Center, Dept of Med/ER Med, New Orleans, Louisiana, United States

REFERENCES:
- [Result] Stryjewski ME, Graham DR, Wilson SE, O'Riordan W, Young D, Lentnek A, Ross DP, Fowler VG, Hopkins A, Friedland HD, Barriere SL, Kitt MM, Corey GR; Assessment of Telavancin in Complicated Skin and Skin-Structure Infections Study. Telavancin versus vancomycin for the treatment of complicated skin and skin-structure infections caused by gram-positive organisms. Clin Infect Dis. 2008 Jun 1;46(11):1683-93. doi: 10.1086/587896. PMID 18444791
- [Result] Wilson SE, O'Riordan W, Hopkins A, Friedland HD, Barriere SL, Kitt MM; ATLAS Investigators. Telavancin versus vancomycin for the treatment of complicated skin and skin-structure infections associated with surgical procedures. Am J Surg. 2009 Jun;197(6):791-6. doi: 10.1016/j.amjsurg.2008.05.012. Epub 2008 Dec 18. PMID 19095213
- [Derived] Stryjewski ME, Barriere SL, O'Riordan W, Dunbar LM, Hopkins A, Genter FC, Corey GR. Efficacy of telavancin in patients with specific types of complicated skin and skin structure infections. J Antimicrob Chemother. 2012 Jun;67(6):1496-502. doi: 10.1093/jac/dks081. Epub 2012 Mar 13. PMID 22416054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: 18 February 2005 to 31 May 2006
Groups:
- Telavancin: Patients with complicated Gram-positive skin and skin structure infections (primarily due to MRSA) were randomized to receive telavancin 10 mg/kg IV once daily. The maximum allowable treatment period was 14 days.
- Vancomycin: Patients with complicated Gram-positive skin and skin structure infections (primarily due to MRSA) were randomized to receive vancomycin 1 Gm every 12 hours. The maximum allowable treatment period was 14 days.
Period: Overall Study
Arm/Group | Telavancin | Vancomycin
Started | 458 | 481
Completed | 425 | 431
Not Completed | 33 | 50
Not completed — Adverse Event | 1 | 5
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 20 | 28
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telavancin | Vancomycin | Total
Number analyzed (Participants) | 458 | 481 | 939
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 377 | 379 | 756
  >=65 years | 81 | 102 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (16.1) | 49.9 (17.0) | 49.5 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 187 | 387
  Male | 258 | 294 | 552
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 84 | 163
  Not Hispanic or Latino | 379 | 397 | 776
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 9 | 16
  Asian | 38 | 44 | 82
  Native Hawaiian or Other Pacific Islander | 4 | 8 | 12
  Black or African American | 69 | 74 | 143
  White | 336 | 343 | 679
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 287 | 310 | 597
  South Africa | 6 | 6 | 12
  Argentina | 35 | 33 | 68
  Canada | 35 | 29 | 64
  Chile | 1 | 2 | 3
  France | 0 | 2 | 2
  Germany | 0 | 4 | 4
  Italy | 2 | 1 | 3
  Korea, Republic of | 14 | 16 | 30
  Lithuania | 12 | 6 | 18
  Peru | 4 | 1 | 5
  Poland | 38 | 43 | 81
  Spain | 2 | 3 | 5
  Taiwan | 20 | 25 | 45
  United Kingdom | 2 | 0 | 2
Diabetes Status [Number; unit: Participants]
  Diabetic | 113 | 118 | 231
  Not diabetic | 345 | 363 | 708

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: The Clinical Response for each patient was determined by the investigator by assessing the patient's clinical signs & symptoms compared with the Baseline evaluation. Cure: resolution of signs and symptoms associated with the skin infection present at study admission such that no further antibiotic therapy was necessary; Not Cured: inadequate response to study therapy; Indeterminate: unable to determine outcome.
Time Frame: 7 to 14 days after the last antibiotic dose
Population: Data for the all-treated population (AT) are presented. The AT and clinically evaluable (CE) populations were considered co-primary.
Measure: Number; unit: patients
Arm/Group | Telavancin | Vancomycin
Number analyzed (Participants) | 458 | 481
patients
  Cure | 358 | 364
  Not cured | 59 | 57
  Indeterminate | 17 | 20
  Missing | 24 | 40
Statistical Analysis 1: Comparison: Telavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 10% was specified based on historical regulatory precedent; 2-sided 95% confidence interval — p-values were not calculated in deference to confidence intervals; 2-sided 95% confidence interval calculated on the difference in cure rates between treatment groups; Risk Difference (RD) = 2.5, 95% CI [-2.9 to 7.9]

ADVERSE EVENTS:
Description: Safety data includes data from all patients treated. Efficacy data does not include data from three sites. Hence, there is a discrepancy between the total numbers of patients in each arm in the safety data vs. the efficacy data.
Arm/Group | Telavancin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 38/503 | 15/509
Other Adverse Events (participants affected / at risk) | 377/503 | 341/509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Telavancin (N=503) | Vancomycin (N=509)
Renal Failure Acute (Renal and urinary disorders) | 3 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 0
Blood creatinine increased (Investigations) | 3 | 0
Drug Hypersensitivity (Immune system disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 0
Renal Insufficiency (Renal and urinary disorders) | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Blood Urea increased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peripheral Occlusive Disease (Vascular disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Abscess Soft Tissue (Infections and infestations) | 1 | 0
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Brain Stem Infarction (Nervous system disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Gangrene (Vascular disorders) | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral Discitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0/503
Non-Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Alanine Aminotransferase increased (Investigations) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Aspartate Aminotransferase increased (Investigations) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Infusion site reaction (General disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1
Rigors (General disorders) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=503) | Vancomycin (N=509)
Anemia (Blood and lymphatic system disorders) | 11 | 10
Abdominal Pain (Gastrointestinal disorders) | 6 | 9
Constipation (Gastrointestinal disorders) | 35 | 24
Diarrhoea (Gastrointestinal disorders) | 36 | 35
Dry Mouth (Gastrointestinal disorders) | 9 | 7
Dyspepsia (Gastrointestinal disorders) | 7 | 7
Loose stools (Gastrointestinal disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 121 | 47
Vomiting (Gastrointestinal disorders) | 49 | 19
Asthenia (General disorders) | 5 | 7
Fatigue (General disorders) | 22 | 10
Infusion site erythema (General disorders) | 17 | 15
Infusion site pain (General disorders) | 20 | 19
Infusion site phlebitis (General disorders) | 12 | 14
Infusion site pruritis (General disorders) | 4 | 9
Infusion site reaction (General disorders) | 7 | 7
Pyrexia (General disorders) | 6 | 2
Rigors (General disorders) | 19 | 7
Drug Hypersensitivity (Immune system disorders) | 5 | 6
Urinary Tract Infection (Infections and infestations) | 13 | 3
Vaginal mycosis (Infections and infestations) | 4 | 6
Alanine Aminotransferase increased (Investigations) | 6 | 13
Aspartate Aminotransferase increased (Investigations) | 6 | 10
Blood Creatinine Increased (Investigations) | 9 | 3
Anorexia (Metabolism and nutrition disorders) | 7 | 1
Decreased appetite (Metabolism and nutrition disorders) | 12 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 9
Dizziness (Nervous system disorders) | 28 | 18
Dysgeusia (Nervous system disorders) | 155 | 31
Headache (Nervous system disorders) | 48 | 51
Hypoaesthesia (Nervous system disorders) | 3 | 6
Paraesthesia (Nervous system disorders) | 3 | 7
Somnolence (Nervous system disorders) | 8 | 3
Anxiety (Psychiatric disorders) | 8 | 8
Insomnia (Psychiatric disorders) | 19 | 33
Renal Failure Acute (Renal and urinary disorders) | 6 | 0
Urine Abnormality (Renal and urinary disorders) | 53 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Erythema (Skin and subcutaneous tissue disorders) | 3 | 6
Pruritis (Skin and subcutaneous tissue disorders) | 29 | 62
Pruritis generalized (Skin and subcutaneous tissue disorders) | 9 | 20
Rash (Skin and subcutaneous tissue disorders) | 18 | 20
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 7
Flushing (Vascular disorders) | 6 | 14
Hypertension (Vascular disorders) | 6 | 6
Hypotension (Vascular disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less